CLINICAL TRIAL: NCT03589573
Title: Effect of Trunk and Lower Extremity Muscle Strength on Hamstring Flexibility in Children With Duchenne Muscular Dystrophy
Brief Title: Effect of Muscle Strength on Hamstring Flexibility in Children With Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Lütfiye AKKURT, Principal investigator, Hacettepe University
Other Study IDs: GO 16/740-1
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Duchenne Muscular Dystrophy; Muscle Strength; Lower Extremity; Hamstring Contractures
Keywords: Duchenne Muscular Dystrophy; muscle strength; hamstring flexibility; back muscle; lower extremity
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigator researched that the effect of trunk and lower extremity muscle strength on hamstring flexibility in children with Duchenne Muscular Dystrophy.

DETAILED DESCRIPTION:
Thirty children were asessed by physical therapist. Nineteen children was Level 1 and eleven children was Level 2 according to Brooke Lower Extremity Functional Classification Scale.

ELIGIBILITY:
Inclusion Criteria:

* Getting a Duchenne Muscular Dystrophy diagnosis,
* Being in ambulatuar phases and independently climbing four stairs
* To be cooperate to physioterapist's directions

Exclusion Criteria:

* Having severe contracture in the lower extremity
* Having undergone surgery in the past 6 months

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Thirty children whose functional levels were in 1 or 2 according to the Brooke Lower Extremity Functional Classification Scale were included in the study. Flexibilities of hamstrings was evaluated by Popliteal Angle Test. Muscle strenght was assessed with manuel muscle strength test and myometer. correlation between the flexibility of hamstrings and muscle strength tests were examined.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
popliteal angle test | 5 minute
  The popliteal angle test was performed to assess hamstring flexibility. The popliteal angle was measured in a supine position and the hip flexed 90°, and fixed by first physical therapist. Opposite knee and hip were placed in extension position. Then, the child was asked to rise lower leg straight. The incomplete angle for full extension of the knee was the popliteal angle.

SECONDARY OUTCOMES:
trunk and lower extremity muscle strength test | 20 minute
  Trunk and lower extremity muscle strength was assessed manual muscle strength and myometer. Any test was performed three times and best value was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfiye Akkurt, Msc., Principal Investigator — Hacettepe University; Öznur Yılmaz, Prof., Study Director — Hacettepe University; İpek Gürbüz, Assoc.Prof., Principal Investigator — Hacettepe University; Ayşe Karaduman, Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No